CLINICAL TRIAL: NCT03726918
Title: Identification of New Predictive Osseointegration Bio-Markers of the Prosthetic Implant in Patients With OsteoArthritis
Acronym: BioPreIOA
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: BioPreIOA
Record Dates: First submitted 2018-09-27; First posted 2018-11-01 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-07

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The isolated cells of synoviocytes, osteoblasts and chondrocytes from tissue samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Osteoarthritis: Surgery for implantation of a prosthesis in case of Osteoarthritis
  Interventions: Procedure: Surgery for implantation of a prosthesis
- Non Osteoarthritis: Surgery for implantation of a prosthesis fon non Osteoarthritis cases
  Interventions: Procedure: Surgery for implantation of a prosthesis

INTERVENTIONS:
Procedure: Surgery for implantation of a prosthesis — Analysis of micro Ribo Nucleic Acid (RNA) expressed by the synoviocytes, osteoblasts and chondrocytes
  Other Names: non-osteoarthritis arm

SUMMARY:
The study involves the isolation and cellular, molecular and proteomic characterization of synoviocytes, osteoblasts and chondrocytes from tissue samples obtained from patients undergoing surgery of endo or arthroplasty for osteoarthritis (Experimental Group) or interventions for other causes such as for example periarticular fracture requiring the implantation of a prosthesis (Control Group)

DETAILED DESCRIPTION:
The study involves the isolation and cellular, molecular and proteomic characterization of synoviocytes, osteoblasts and chondrocytes from tissue samples obtained from patients undergoing surgery of endo or arthroplasty for osteoarthritis (Experimental Group) or interventions for other causes such as for example periarticular fracture requiring the implantation of a prosthesis (Control Group) Deeper analysis of micro Ribo Nucleic Acid (RNA) and Non Coding RNA expressed by the synoviocytes, osteoblasts and chondrocytes will be performed in order to understand their possible involvement in pathways of osteogenic differentiation, through suitable experimental in vitro models of co-cultures. In particular, investigators will focus on the cross-talk between synoviocytes and osteoblasts, cell populations involved in the post-surgical articular microenvironment and on which the osteointegration process of the joint prosthesis depends.

ELIGIBILITY:
Inclusion Criteria:

1. Male and Female patients > 40 years old hospitalized for surgery of endo- or arthroplasty for Osteoarthritis or for surgery for joint traumatic diseases (eg femoral neck fractures) requiring the implantation of a prosthesis
2. Interval of at least three months from any previous infiltrative treatment of any kind;
3. Patients able to provide written informed consent to the study.

Exclusion Criteria:

1. Severe cognitive defects or psychiatric disorders;
2. Tumor pathologies or concurrent antineoplastic therapies;
3. Autoimmune diseases (rheumatoid arthritis);
4. Surgery that involves the joint

Min Age: 40 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Male and female patients of age >40 years undergoing surgery of endo or arthroplasty for osteoarthritis or ifor other causes requiring the implantation of a prosthesis
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2018-12-14 (Actual); Primary Completion 2020-06-20 (Actual); Study Completion 2020-06-20 (Actual)

PRIMARY OUTCOMES:
miRNAs and LncRNA | at the time of surgery (Day0)
  expression of miRNAs and LncRNA, from synoviocytes, osteoblasts and chondrocytes detected at the time of surgery

SECONDARY OUTCOMES:
Biomarkers useful for predicting the efficiency of osseointegration of the implant | at the time of surgery (Day0)
  the mRNAs and the identified proteins will be analyzed through the use of specific software, such as TargetScanPrediction.
Validation of data obtained on miRNAs and lncRNAs | at the time of surgery (Day0)
  Through in vitro co-culture systems, investigators will evaluate the role of previously identified miRNAs and lncRNAs in cross-talk between osteoblasts and synoviocytes isolated from patients with osteoarthritis.

CONTACTS AND LOCATIONS:
Overall Officials: Gianluca Giavaresi, MD, Study Chair — Isituto Ortopedico Rizzoli
Locations (1):
- IRCCS Istituto Ortopedico Rizzoli, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: No
No Individual Patient Data sharing plan has been implemented

REFERENCES:
- [Background] Costa V, Raimondi L, Conigliaro A, Salamanna F, Carina V, De Luca A, Bellavia D, Alessandro R, Fini M, Giavaresi G. Hypoxia-inducible factor 1Alpha may regulate the commitment of mesenchymal stromal cells toward angio-osteogenesis by mirna-675-5P. Cytotherapy. 2017 Dec;19(12):1412-1425. doi: 10.1016/j.jcyt.2017.09.007. Epub 2017 Oct 27. PMID 29111380
- [Background] Pelletier JP, Martel-Pelletier J, Abramson SB. Osteoarthritis, an inflammatory disease: potential implication for the selection of new therapeutic targets. Arthritis Rheum. 2001 Jun;44(6):1237-47. doi: 10.1002/1529-0131(200106)44:63.0.CO;2-F. No abstract available. PMID 11407681
- [Background] Marijnissen AC, Lafeber FP. Re: E. B. Hunziker. Articular cartilage repair: basic science and clinical progress. A review of the current status and prospects. Osteoarthritis and Cartilage 2002; 10:432-63. Osteoarthritis Cartilage. 2003 Apr;11(4):300-1; author reply 302-4. doi: 10.1016/s1063-4584(02)00346-1. No abstract available. PMID 12681957
- [Background] Zhang M, Lygrisse K, Wang J. Role of MicroRNA in Osteoarthritis. J Arthritis. 2017 Apr;6(2):239. doi: 10.4172/2167-7921.1000239. Epub 2017 Apr 28. PMID 28758052

DOCUMENTS (1):
  • Study Protocol (2018-04-24): https://cdn.clinicaltrials.gov/large-docs/18/NCT03726918/Prot_000.pdf